CLINICAL TRIAL: NCT02408939
Title: Effect of Stress-dose Steroids on Post-resuscitation Infectious (Septic) Complications After In-hospital Cardiac Arrest. Individual Patient Data-based Re-analysis of Synthesized Prior Randomized Clinical Trial Data
Brief Title: Steroids and Post-resuscitation Infectious (Septic) Complications
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Spyros D. Mentzelopoulos, Associate Professor in Intensive Care Medicine, University of Athens
Other Study IDs: 14/9/1/2015 IPDRA
Record Dates: First submitted 2015-03-27; First posted 2015-04-06 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2017-03

CONDITIONS: Infections; Cardiac Arrest
MeSH Terms: conditions — Infections; Heart Arrest

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention: Patients resuscitated from in-hospital cardiac arrest and treated with stress-dose hydrocortisone for postresuscitation shock
  Interventions: Drug: Stress-dose hydrocortisone
- Control: Patients resuscitated from in-hospital cardiac arrest and treated according to contemporary standards that did not include stress-dose steroids for postresuscitation shock

INTERVENTIONS:
Drug: Stress-dose hydrocortisone — Patients with postresuscitation shock received stress-dose (300 mg) of hydrocortisone for 7 days maximum followed by gradual taper and discontinuation over 48 hours after either the resolution of their hemodynamic instability or day 7 of treatment.
  Other Names: Solucortef
  Groups: Intervention

SUMMARY:
Postresuscitation disease is characterized by post-insult systemic inflammation, adrenal insufficiency, and circulatory failure. Such severe pathology may be associated with increased susceptibility to infectious complications and increased risk of death due to postresuscitation septic shock. The latter may be attenuated by stress-dose steroids. In this re-analysis of synthesized randomized clinical trial (RCT) data, the investigators will use individual patient data from two prior RCTs of in-hospital cardiac arrest (NCT00411879 & NCT00729794), in order to determine the effect of stress-dose steroids on the severity of postresuscitation infectious complications, and more specifically, on the risk of septic shock-associated death.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Patients successfully resuscitated after cardiac arrest experience a "sepsis-like" syndrome characterized by cytokine storm, endotoxemia, coagulopathy, and various degrees of adrenal insufficiency. These pathophysiological mechanisms contribute to the development of circulatory failure, i.e. post-resuscitation shock. Post-resuscitation shock patients resuscitated from vasopressor-requiring cardiac arrest are frequently poorly responsive to high-rate vasopressor infusions (e.g. norepinephrine ≥0.5 μg/kg/min) and intravenous fluids.

The postresuscitation systemic inflammatory response syndrome (SIRS) may be partly caused and subsequently amplified by ischemia/reperfusion (I/R)-associated disruption of the intestinal mucosal barrier. Steroids may suppress key events of I/R injury propagation. Furthermore, in shock states, stress-dose steroids improve vascular responsiveness to vasopressors and preserve monocyte and neutrophil phagocytosis, and dendritic cell function. Low-dose steroids may reduce the mortality of severely ill patients with septic shock.

Nosocomial infections constitute an important cause of postresuscitation mortality. We hypothesized that exposure to stress-dose steroids during and/or after CPR may be associated with reduced risk of death due to postresuscitation infectious complications. To test this hypothesis, we combined data from two prior, prospective studies of in-hospital cardiac arrest. These studies compared the combination of vasopressin, steroids, and epinephrine (VSE) to epinephrine alone, with respect to survival to hospital discharge and good functional outcome. Patients with post-resuscitation shock of the VSE groups received stress dose hydrocortisone (300 mg/day for 7 days maximum, followed by gradual taper at a rate of 100 mg / day and discontinuation on day 10). Patients with post-resuscitation shock of the control groups received saline placebo. Follow-up rates were high in both studies and the reported incidence of post-resuscitation infectious complications was similar in the VSE and control groups.

METHODS Study Design Retrospective analysis of prospectively collected data from two randomized, clinical studies. Study participants were hospitalized in intensive or coronary care units (ICUs or CCUs) of three tertiary care centers: Evaggelismos General Hospital and 401 Greek Army Hospital (both in Athens, Greece), and University Hospital of Larissa, Larissa, Greece.

Ethics and Approval The present analysis is not associated with any clinical intervention, and therefore, the investigators have applied for a waiver of informed consent from either the patient or his/her next of kin. Moreover, the investigators have requested the permission to confirm previously recorded microbiological data through the hospitals' electronic databases The institutional review boards (IRBs) of the aforementioned hospitals have granted their approval for the current study. Evaggelismos Hospital approval No. 14/9/1/2015; 401 Greek Army Hospital approval No. 3/2015/5/2/2015; Larissa University Hospital approval No. 58905/2014/14/1/2015. Modifications of statistical terminology [from individual patient data (IPD) meta-analysis to IPD re-analysis] and of infections' classification in the definition of the primary outcome were also approved by the Evaggelismos IRB (respective Approval Nos. 30/25/2/2016 and 29/25/2/2016) and communicated to the other 2, aforementioned IRBs. These approvals were ratified by the IRBs of the other 2 participating centers (401 Greek Army Hospital, IRB Decision No.: 4-2016/6/4/2016; Larissa University Hospital, IRB Decision No.: 5/19-5-2016/Θ.18). Additional, significant amendments of the analysis protocol aimed at primarily evaluating the effect of stress-dose steroids on lethal septic shock were approved by the Evaggelismos IRB (Approval No. 9/26/1/2017) and appropriately communicated to the other 2, aforementioned IRBs.

Analysis Endpoints are presented in the dedicated subsection. Patients The reference study population consists of 368 patients (Evaggelismos Hospital, n=288/368=78.2%) with in-hospital cardiac arrest, who required epinephrine during cardiopulmonary resuscitation (CPR) according to the 2005 Guidelines for Resuscitation. During CPR, VSE group patients (n=178) also received vasopressin and methylprednisolone and controls (n=190) the respective saline placebos. At 4 hours after CPR, there were 211 surviving patients (VSE group, n=115), who were evaluated for postresuscitation shock. One hundred three VSE group patients were then assigned to stress-dose hydrocortisone and 88 controls to saline placebo. One hundred two VSE group patients and 15 controls were actually treated with stress-dose hydrocortisone (n=117). One VSE group patient did not receive stress dose hydrocortisone due to pharmacist error; however, the patient did receive 40 mg of methylprednisolone during CPR.

Definitions Essential prerequisites for the applicability of the below-provided definitions of infections to determine their (prior) occurence in the participants of the included studies will include the presence of confirmatory investigator recordings (for the prior diagnoses of these infections) and also the retrieval of confirmatory microbiological data from hospital records.

Ventilator-associated pneumonia (VAP) will be defined as new (or worsening if already present) chest x-ray infiltrate and at least 2 of the following 3 findings: worsening of respiratory secretions (to purulent or muco-purulent), leucocytosis or leucopenia (>11000/μL or <4000/μL respectively), and fever or hypothermia (>38 degrees Celcius or <36 degrees Celcius respectively). VAP diagnosis will require at least 48 hours of postresuscitation endotracheal intubation and mechanical ventilation. VAP will be confirmed by a positive tracheobronchial aspirate sample with ≥1000000 Colony Forming Units (CFUs)/μL] and / or a concurrent blood culture positive for the same pathogen.

Ventilator-associated tracheobronchitis (VAT) will be defined as fever (>38 degrees Celcius) not attributable to another infectious complication and positive tracheobronchial aspirate culture (with ≥1000000 CFUs/μL) yielding a new bacteria (not present at intubation), and no radiographic signs of new pneumonia.

Bacteremia (or Fungemia) will be defined as isolation of a pathogen from at least one blood culture set (in cases of coagulase negative Staphylococcus species, or Corynebacterium species, 2 positive blood culture sets will be required). Septic shock will be defined as bacteremia / fungemia plus circulatory failure with at least 30% increase in norepinephrine infusion requirements after day 3 postarrest.

Urinary tract infection will be defined as fever or hypothermia and presence of at least one pathogen in a urine sample culture at a concentration of ≥100000 CFUs/μL.

Post-resuscitation shock, organ / system failures, acute respiratory distress syndrome, hyperglycemia, and survival to hospital discharge with good functional outcome will be defined as in the 2 included VSE studies. Organ failure free days and ventilator free days will be determined as in the 2 included VSE studies.

Statistical Analysis Plan All analyses will be performed with the Statistical Package for Social Sciences version 22.0 (IBM, Armonk, NY, USA). As this is not a randomized study, patient baseline characteristics will be compared between the Steroids and No Steroids groups. Distribution normality will be tested by Kolmogorov-Smirnov test. Dichotomous and categorical variables will be compared by a two-sided chi-square or Fisher's exact test. Continuous variables will be compared by a two-tailed, independent samples t test or Mann-Whitney exact U test.

We will conduct a cumulative incidence competing risks analysis (CICR) to determine cause-specific hazard ratios (CSHRs) and their 95% confidence intervals (CIs) for death due to a postresuscitation infection, i.e., lethal septic shock, death due to a noninfectious cause, and poor inhospital outcome (as defined in the outcome measures subsection).

Prespecified risk factors for physical death or poor inhospital outcome will be group (Intervention vs. Control); cardiac arrest cause (cardiac vs. non-cardiac); cardiac arrest area (monitored vs. non-monitored), initial cardiac arrest rhythm (shockable vs. non-shockable); cardiac arrest time (i.e. weekday vs. holiday and nighttime vs. morning-to-late evening), advanced life support (ALS)-related bicarbonate dose; time from resuscitation team call to ALS initiation plus ALS duration; and therapeutic hypothermia (yes vs. no).

Additional analyses will include addition of early postresuscitation mean arterial pressure as covariate to the multivariable CICR Cox models

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with refractory inhospital cardiac arrest, defined as epinephrine requirement for ventricular fibrillation/tachycardia or asystole/pulseless electrical activity according to guidelines for resuscitation 2005

Exclusion Criteria:

* Age < 18 years
* Terminal illness or do-not resuscitate status
* Cardiac arrest due to exsanguination
* Cardiac arrest before hospital admission
* Pre-arrest treatment with intravenous corticosteroids
* Previous enrollment in or exclusion from the 2 studies included in the re-analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with vasopressor-requiring, inhospital cardiac arrest, i.e., with asystole, pulseless electrical activity, or ventricular fibrillation/pulseless ventricular tachycardia not responsive to two attempts at defibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Lethal septic shock due to a postresuscitation infection. | Post-resuscitation length of ICU / CCU stay [60 days].
  Septic shock associated with microbiologically confirmed ventilator-associated pneumonia (VAP), ventilator-associated tracheobronchitis (VAT), central venous catheter-related bloodstream infection, bacteremia/fungemia of presumed extrapulmonary origin, urinary tract infection, and "other" infections (e.g. endocarditis, soft tissue infection, viral infection).

SECONDARY OUTCOMES:
Organ failure-free days | Post-resuscitation length of ICU / CCU stay [60 days].
  Organ failure-free days: Numbers of days without circulatory, respiratory, renal, hepatic, coagulation, or neurologic failure.
Ventilator-free days | Post-resuscitation length of ICU / CCU stay [60 days].
  Number of days with sustained spontaneous breathing
Non-infectious complications of stress-dose corticosteroid treatment | Post-resuscitation length of ICU / CCU stay [60 days].
  Hyperglycemia, peptic ulcer bleeding, and neuromuscular weakness
Death due to noninfectious causes | Post-resuscitation length of ICU / CCU stay [60 days].
  Death of any cause besides a postresuscitation infectious complicaiton
Poor inhospital outcome | Post-resuscitation length of ICU / CCU stay [60 days].
  Physical death during patient follow-up or postresuscitation neurologic failure [i.e. Glasgow Coma Score (GCS) ≤9 while being circulatory failure-free and ≥24 h sedation-free] that was associated with a Cerebral Performance Category score of ≥3 at the end of the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Spyros D Mentzelopoulos, MD, PhD, Principal Investigator — University of Athens Medical School; Spyros D Mentzelopoulos, MD, PhD, Study Director — University of Athens Medical School; Spyros G Zakynthinos, MD, PhD, Study Chair — University of Athens Medical School
Locations (5):
- Service d'anesthésie et des réanimations chirurgicales, ôHôpitaux Universitaires Henri Mondor, Assistance Publique des Hôpitaux de Paris, Université Paris Est, Faculté de Médecine, Créteil, France
- Greece (4):
  - Department of Intensive Care Medicine, Evaggelismos Hospital, Athens, Attica
  - 401 General Military Hospital of Athens, Athens, Attica
  - University General Hospital of Larissa, Larissa, Thessaly
  - President Hellenic Society of Cardiopulmonary Resuscitation, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adrie C, Adib-Conquy M, Laurent I, Monchi M, Vinsonneau C, Fitting C, Fraisse F, Dinh-Xuan AT, Carli P, Spaulding C, Dhainaut JF, Cavaillon JM. Successful cardiopulmonary resuscitation after cardiac arrest as a "sepsis-like" syndrome. Circulation. 2002 Jul 30;106(5):562-8. doi: 10.1161/01.cir.0000023891.80661.ad. PMID 12147537
- [Background] Adrie C, Laurent I, Monchi M, Cariou A, Dhainaou JF, Spaulding C. Postresuscitation disease after cardiac arrest: a sepsis-like syndrome? Curr Opin Crit Care. 2004 Jun;10(3):208-12. doi: 10.1097/01.ccx.0000126090.06275.fe. PMID 15166838
- [Background] Pene F, Hyvernat H, Mallet V, Cariou A, Carli P, Spaulding C, Dugue MA, Mira JP. Prognostic value of relative adrenal insufficiency after out-of-hospital cardiac arrest. Intensive Care Med. 2005 May;31(5):627-33. doi: 10.1007/s00134-005-2603-7. Epub 2005 Apr 19. PMID 15838680
- [Background] Kim JJ, Lim YS, Shin JH, Yang HJ, Kim JK, Hyun SY, Rhoo I, Hwang SY, Lee G. Relative adrenal insufficiency after cardiac arrest: impact on postresuscitation disease outcome. Am J Emerg Med. 2006 Oct;24(6):684-8. doi: 10.1016/j.ajem.2006.02.017. PMID 16984836
- [Background] Hekimian G, Baugnon T, Thuong M, Monchi M, Dabbane H, Jaby D, Rhaoui A, Laurent I, Moret G, Fraisse F, Adrie C. Cortisol levels and adrenal reserve after successful cardiac arrest resuscitation. Shock. 2004 Aug;22(2):116-9. doi: 10.1097/01.shk.0000132489.79498.c7. PMID 15257083
- [Background] Tsai MS, Huang CH, Chang WT, Chen WJ, Hsu CY, Hsieh CC, Yang CW, Chiang WC, Ma MH, Chen SC. The effect of hydrocortisone on the outcome of out-of-hospital cardiac arrest patients: a pilot study. Am J Emerg Med. 2007 Mar;25(3):318-25. doi: 10.1016/j.ajem.2006.12.007. PMID 17349907
- [Background] Schultz CH, Rivers EP, Feldkamp CS, Goad EG, Smithline HA, Martin GB, Fath JJ, Wortsman J, Nowak RM. A characterization of hypothalamic-pituitary-adrenal axis function during and after human cardiac arrest. Crit Care Med. 1993 Sep;21(9):1339-47. doi: 10.1097/00003246-199309000-00018. PMID 8396524
- [Background] Nolan JP, Deakin CD, Soar J, Bottiger BW, Smith G; European Resuscitation Council. European Resuscitation Council guidelines for resuscitation 2005. Section 4. Adult advanced life support. Resuscitation. 2005 Dec;67 Suppl 1:S39-86. doi: 10.1016/j.resuscitation.2005.10.009. No abstract available. PMID 16321716
- [Background] Keh D, Boehnke T, Weber-Cartens S, Schulz C, Ahlers O, Bercker S, Volk HD, Doecke WD, Falke KJ, Gerlach H. Immunologic and hemodynamic effects of "low-dose" hydrocortisone in septic shock: a double-blind, randomized, placebo-controlled, crossover study. Am J Respir Crit Care Med. 2003 Feb 15;167(4):512-20. doi: 10.1164/rccm.200205-446OC. Epub 2002 Nov 8. PMID 12426230
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Mermel LA, Allon M, Bouza E, Craven DE, Flynn P, O'Grady NP, Raad II, Rijnders BJ, Sherertz RJ, Warren DK. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jul 1;49(1):1-45. doi: 10.1086/599376. PMID 19489710
- [Background] Hooton TM, Bradley SF, Cardenas DD, Colgan R, Geerlings SE, Rice JC, Saint S, Schaeffer AJ, Tambayh PA, Tenke P, Nicolle LE; Infectious Diseases Society of America. Diagnosis, prevention, and treatment of catheter-associated urinary tract infection in adults: 2009 International Clinical Practice Guidelines from the Infectious Diseases Society of America. Clin Infect Dis. 2010 Mar 1;50(5):625-63. doi: 10.1086/650482. PMID 20175247
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] A randomized clinical trial of calcium entry blocker administration to comatose survivors of cardiac arrest. Design, methods, and patient characteristics. The Brain Resuscitation Clinical Trial II Study Group. Control Clin Trials. 1991 Aug;12(4):525-45. doi: 10.1016/0197-2456(91)90011-a. PMID 1657528
- [Background] Vollmar B, Menger MD. Intestinal ischemia/reperfusion: microcirculatory pathology and functional consequences. Langenbecks Arch Surg. 2011 Jan;396(1):13-29. doi: 10.1007/s00423-010-0727-x. Epub 2010 Nov 19. PMID 21088974
- [Background] Davies KJ, Walters JH, Kerslake IM, Greenwood R, Thomas MJ. Early antibiotics improve survival following out-of hospital cardiac arrest. Resuscitation. 2013 May;84(5):616-9. doi: 10.1016/j.resuscitation.2012.11.004. Epub 2012 Nov 12. PMID 23153650
- [Background] Chalkias A, Scheetz MH, Gulati A, Xanthos T. Periarrest intestinal bacterial translocation and resuscitation outcome. J Crit Care. 2016 Feb;31(1):217-20. doi: 10.1016/j.jcrc.2015.09.015. Epub 2015 Sep 25. PMID 26481507
- [Background] Haller B, Schmidt G, Ulm K. Applying competing risks regression models: an overview. Lifetime Data Anal. 2013 Jan;19(1):33-58. doi: 10.1007/s10985-012-9230-8. Epub 2012 Sep 26. PMID 23010807
- [Background] Trzeciak S, Jones AE, Kilgannon JH, Milcarek B, Hunter K, Shapiro NI, Hollenberg SM, Dellinger P, Parrillo JE. Significance of arterial hypotension after resuscitation from cardiac arrest. Crit Care Med. 2009 Nov;37(11):2895-903; quiz 2904. doi: 10.1097/ccm.0b013e3181b01d8c. PMID 19866506
- [Background] Tsai MS, Chuang PY, Yu PH, Huang CH, Tang CH, Chang WT, Chen WJ. Glucocorticoid use during cardiopulmonary resuscitation may be beneficial for cardiac arrest. Int J Cardiol. 2016 Nov 1;222:629-635. doi: 10.1016/j.ijcard.2016.08.017. Epub 2016 Aug 4. PMID 27517652
- [Background] Callaway CW, Soar J, Aibiki M, Bottiger BW, Brooks SC, Deakin CD, Donnino MW, Drajer S, Kloeck W, Morley PT, Morrison LJ, Neumar RW, Nicholson TC, Nolan JP, Okada K, O'Neil BJ, Paiva EF, Parr MJ, Wang TL, Witt J; Advanced Life Support Chapter Collaborators. Part 4: Advanced Life Support: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2015 Oct 20;132(16 Suppl 1):S84-145. doi: 10.1161/CIR.0000000000000273. No abstract available. PMID 26472860
- [Result] Mentzelopoulos SD, Zakynthinos SG, Tzoufi M, Katsios N, Papastylianou A, Gkisioti S, Stathopoulos A, Kollintza A, Stamataki E, Roussos C. Vasopressin, epinephrine, and corticosteroids for in-hospital cardiac arrest. Arch Intern Med. 2009 Jan 12;169(1):15-24. doi: 10.1001/archinternmed.2008.509. PMID 19139319
- [Result] Mentzelopoulos SD, Malachias S, Chamos C, Konstantopoulos D, Ntaidou T, Papastylianou A, Kolliantzaki I, Theodoridi M, Ischaki H, Makris D, Zakynthinos E, Zintzaras E, Sourlas S, Aloizos S, Zakynthinos SG. Vasopressin, steroids, and epinephrine and neurologically favorable survival after in-hospital cardiac arrest: a randomized clinical trial. JAMA. 2013 Jul 17;310(3):270-9. doi: 10.1001/jama.2013.7832. PMID 23860985
- [Derived] Mentzelopoulos SD, Mongardon N, Xanthos T, Zakynthinos SG. Possible significance of hemodynamic and immunomodulatory effects of early stress-dose steroids in cardiac arrest. Crit Care. 2016 Jul 20;20(1):211. doi: 10.1186/s13054-016-1384-4. No abstract available. PMID 27436285